CLINICAL TRIAL: NCT05810285
Title: Total Knee Arthroplasty With Vitamin E Polyethylene
Status: Completed | Type: Observational
Sponsor: Permedica spa (Industry)
Responsible Party: Sponsor
Other Study IDs: VITALECOQ2020
Record Dates: First submitted 2023-03-28; First posted 2023-04-12 (Actual); Results first posted 2024-12-06 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-10

CONDITIONS: Knee Osteoarthritis
Keywords: total knee arthroplasty; vitamin E; polyethylene; aseptic loosening; osteolysis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteolysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- VITAMIN E: Patients who received cemented total knee arthroplasty with vitamin E blended polyethylene mobile bearing
  Interventions: Device: GKS Prime Flex Mobile knee
- POLYETHYLENE: Patients who received cemented total knee arthroplasty with conventional polyethylene mobile bearing
  Interventions: Device: GKS Prime Flex Mobile knee

INTERVENTIONS:
Device: GKS Prime Flex Mobile knee — Total knee arthroplasty with a cemented mobile bearing bicompartmental knee prosthesis

SUMMARY:
The aim of this observational study is to investigate if there is any difference in survival rate, clinical and radiological results after total knee replacement with vitamin E-blended polyethylene in comparison to conventional polyethylene at minimum 7-year follow-up

ELIGIBILITY:
Inclusion Criteria:

* Patient who received primary cemented total knee arthroplasty with GKS Prime Flex Mobile knee by Permedica Orthopaedics with vitamin E polyethylene bearing or with conventional polyethylene bearing.
* Minimum 7-year follow-up;
* Age ≥ 18 and < 85 years;
* Patient who signed informed consent.

Exclusion Criteria:

* Patient who received primary cemented total knee arthroplasty with a different knee prosthetic design;
* Patient already enrolled in other clinical studies.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received primary cemented total knee arthroplasty with GKS Prime Flex Mobile knee by Permedica Orthopaedics with vitamin E polyethylene bearing or with conventional polyethylene bearing
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Spezia, MD, Principal Investigator — Ospedale Centro Ortopedico di Quadrante
Locations (1):
- Ospedale Centro Ortopedico di Quadrante, Omegna, Verbania, Italy

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During recruitment process, 350 total knee arthroplasties (181 with vitamin E polyethylene and 169 with conventional polyethylene) were identified as eligible. Overall 151 total knee arthroplasties were lost to follow-up and were not enrolled (79 with vitamin E polyethylene and 72 with conventional polyethylene). 186 participants (199 knees) were enrolled.
Pre-assignment Details: 186 participants (199 knees) were enrolled in the study and were assigned to each arm
Units Other Than Participants: Knees (knee implants)
Groups:
- VITAMIN E: Cemented total knee arthroplasty with vitamin E blended polyethylene mobile bearing and GKS Prime Flex Mobile knee
- POLYETHYLENE: Cemented total knee arthroplasty with conventional polyethylene mobile bearing and GKS Prime Flex Mobile knee
Period: Overall Study
Arm/Group | VITAMIN E | POLYETHYLENE
Started | 95; 102 Knees (knee implants) | 91; 97 Knees (knee implants)
Completed | 73; 80 Knees (knee implants) | 54; 60 Knees (knee implants)
Not Completed | 22; 22 Knees (knee implants) | 37; 37 Knees (knee implants)
Not completed — Death | 4 | 21
Not completed — Adverse Event | 18 | 16

BASELINE CHARACTERISTICS:
Population: Baseline Analysis Population included overall number of implants (knees) without those implants lost to follow-up. Patients deceased of causes unrelated to their implant with no history of implant revision, as documented by medical records and by telephone contact with their family, will be included and considered as censored events in survival analysis
Units Other Than Participants: Knees (Knee implants)
Groups:
- Total: Total of all reporting groups
Arm/Group | VITAMIN E | POLYETHYLENE | Total
Number analyzed (Participants) | 95 | 91 | 186
Number analyzed (Knees (Knee implants)) | 102 | 97 | 199
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (6.7) | 75.3 (5.7) | 70.1 (7.9)
Sex: Female, Male [Count of Units; unit: Knees (Knee implants)]
  Female | 61 | 80 | 141
  Male | 41 | 17 | 58
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0
Follow-up [Mean (Standard Deviation); unit: years] | 8.5 (2.1) | 8.3 (2.2) | 8.4 (2.1)
Diagnosis [Count of Units; unit: Knees (Knee implants)]
  Osteoarthritis | 98 | 96 | 194
  Rheumatoid arthritis | 2 | 0 | 2
  Post-traumatic osteoarthritis | 2 | 1 | 3
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.9 (5.9) | 27.8 (5.1) | 29.0 (5.6)

OUTCOME MEASURES:

1. Primary Outcome: Implant Survival for Aseptic Loosening
Description: Kaplan-Meier cumulative survival with revision due to aseptic loosening as the end-point
Time Frame: 10-year follow-up
Measure: Number (95% Confidence Interval); unit: percentage of survival implants
Units Other Than Participants: Knees (knee implants)
Arm/Group | VITAMIN E | POLYETHYLENE
Number analyzed (Participants) | 95 | 91
Number analyzed (Knees (knee implants)) | 102 | 97
percentage of survival implants | 95.0 [88.5 to 97.8] | 97.8 [91.6 to 99.4]

2. Secondary Outcome: Implant Survival for Any Reason
Description: Kaplan-Meier cumulative survival with revision due to any reason as the end-point
Time Frame: 10-year follow-up
Measure: Number (95% Confidence Interval); unit: percentage of survival implants
Units Other Than Participants: Knees (knee implants)
Arm/Group | VITAMIN E | POLYETHYLENE
Number analyzed (Participants) | 95 | 91
Number analyzed (Knees (knee implants)) | 102 | 97
percentage of survival implants | 87.6 [75.8 to 93.8] | 89.6 [81.6 to 94.2]

3. Secondary Outcome: Forgotten Joint Score (FJS-12)
Description: Patient related outcome measurement scored from 0 to 100 (higher scores mean better outcomes)
Time Frame: At mean follow-up of 8.5 years and 8.3 years for Vitamin E and Polyethylene, respectively
Population: Number of knees of patients who was contacted by phone or who returned back to hospital for clinical examination follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Knees (knee implants)
Arm/Group | VITAMIN E | POLYETHYLENE
Number analyzed (Participants) | 73 | 54
Number analyzed (Knees (knee implants)) | 80 | 60
score on a scale | 59 (30) | 56 (27)

4. Secondary Outcome: American Knee Society Score (KSS)
Description: Clinical and Functional scores of the knee. Both scores are scored from 0 to 100 (higher scores mean better outcomes)
Time Frame: At mean follow-up of 8.5 years and 8.3 years for Vitamin E and Polyethylene, respectively
Population: Knees of patients who returned back to the hospital for complete clinical and radiographic follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Knees (knee implants)
Arm/Group | VITAMIN E | POLYETHYLENE
Number analyzed (Participants) | 48 | 28
Number analyzed (Knees (knee implants)) | 52 | 31
score on a scale
  KSS - Knee score | 84 (16) | 80 (16)
  KSS - Function score | 77 (26) | 63 (31)

5. Secondary Outcome: Periprosthetic Radiolucent Line
Description: Radiographic sign of bone remodelling around the implant
Time Frame: At mean follow-up of 8.5 years and 8.3 years for Vitamin E and Polyethylene, respectively
Population: Knees of patients who returned back to hospital for clinical and radiographic follow-up.
Measure: Count of Units; unit: Knees (knee implants)
Units Other Than Participants: Knees (knee implants)
Arm/Group | VITAMIN E | POLYETHYLENE
Number analyzed (Participants) | 48 | 28
Number analyzed (Knees (knee implants)) | 52 | 31
Knees (knee implants) | 28 | 10

6. Secondary Outcome: Periprosthetic Osteolysis
Description: Radiographic sign of focal bone resorption around the implant
Time Frame: At mean follow-up of 8.5 years and 8.3 years for Vitamin E and Polyethylene, respectively
Population: Knees of patients who returned back to hospital for clinical and radiographic follow-up
Measure: Count of Units; unit: Knees (knee implants)
Units Other Than Participants: Knees (knee implants)
Arm/Group | VITAMIN E | POLYETHYLENE
Number analyzed (Participants) | 48 | 28
Number analyzed (Knees (knee implants)) | 52 | 31
Knees (knee implants) | 1 | 1

ADVERSE EVENTS:
Time Frame: At mean follow-up of 8.5 years and 8.3 years for Vitamin E and Polyethylene, respectively
Description: Surgical implant revision with prosthetic component replacement and surgical reintervention fall within the Serious adverse events definition
Arm/Group | VITAMIN E | POLYETHYLENE
All-Cause Mortality (participants affected / at risk) | 4/102 | 21/97
Serious Adverse Events (participants affected / at risk) | 18/102 | 16/97
Other Adverse Events (participants affected / at risk) | 22/102 | 14/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VITAMIN E (N=102) | POLYETHYLENE (N=97)
Revision for aseptic loosening (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2)
Revision for any reason other than aseptic loosening (Musculoskeletal and connective tissue disorders) | 5 (5) | 8 (8)
Reintervention for patella resurfacing (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Reintervention for other reason than patella resurfacing (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Deep venous thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardis (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VITAMIN E (N=102) | POLYETHYLENE (N=97)
Stiffness (Musculoskeletal and connective tissue disorders) | 15 (15) | 4 (4)
Painfull knee (Musculoskeletal and connective tissue disorders) | 6 (6) | 6 (6)
Intraoperative bone fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Delayed wound healing (Infections and infestations) | 0 (0) | 2 (2)
Instability (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Higher than expected number of knees lost to follow-up. Non homogeneous groups for age, gender, and BMI, which might have biased results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/85/NCT05810285/Prot_SAP_000.pdf